CLINICAL TRIAL: NCT03066609
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Study of Subcutaneous Secukinumab, to Demonstrate Efficacy After Twelve Weeks of Treatment and to Assess Safety, Tolerability and Long-term Efficacy up to One Year in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis With or Without Psoriatic Arthritis Comorbidity
Brief Title: Study of Efficacy and Safety of Secukinumab in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2318
Record Dates: First submitted 2017-02-22; First posted 2017-02-28 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis; Secukinumab; Skin condition; skin disease; itching; psoriasis vulgaris; immune-mediated systemic disease; skin lesions; scaly patches; papules; psoriasis
MeSH Terms: conditions — Skin Diseases; Pruritus; Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Secukinumab 150mg (Experimental): Secukinumab 150mg s.c.
  Interventions: Drug: Secukinumab 150 mg s.c.
- Secukinumab 300mg (Experimental): Secukinumab 300mg s.c.
  Interventions: Drug: Secukinumab 300 mg s.c.
- Placebo (Placebo Comparator): Placebo to secukinumab s.c
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab 150 mg s.c. — 150 mg s.c. at randomization, Weeks 1, 2, 3, 4 and every 4 weeks till Week 48
  Arms: Secukinumab 150mg
Drug: Secukinumab 300 mg s.c. — 300 mg s.c. at randomization, Weeks 1, 2, 3, 4 and every 4 weeks till Week 48
  Arms: Secukinumab 300mg
Drug: Placebo — Placebo 150 or 300 mg s.c at randomization, Weeks 1, 2, 3, 4, and 8. PASI responders at week 12 continued to receive placebo till Week 48. PASI non-responders at Week 12 received Secukinumab 300mg at Weeks 12, 13, 14, 15, 16 and every 4 weeks till Week 48
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine if secukinumab is effective and safe in the treatment of plaque type psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give a written, signed and dated informed consent.
2. Men or women at least 18 years of age at time of screening.
3. Chronic plaque-type psoriasis present for at least 6 months and diagnosed before Baseline.
4. Moderate to severe psoriasis as defined at Baseline by:

   * PASI score of 12 or greater, and
   * IGA mod 2011 score of 3 or greater (based on a static scale of 0 - 4), and
   * Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
5. Candidate for systemic therapy. This is defined as a subject having moderate to severe chronic plaque-type psoriasis that is inadequately controlled by

   * topical treatment and/or,
   * phototherapy and/or,
   * previous systemic therapy.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Baseline.
2. Drug-induced psoriasis.
3. Ongoing use of prohibited treatments.
4. Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL-17 or the IL-17 receptor.
5. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- China (13):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xicheng Direct, Beijing Municipality
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Hungary (3):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Orosháza
- Malaysia (2):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Batu Caves
- Philippines (2):
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Quezon City
- Thailand (2):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Manisa
  - Novartis Investigative Site, Mersin

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cai L, Zhang JZ, Yao X, Gu J, Liu QZ, Zheng M, Zhang SF, Xu JH, Li CX, Cheng H, Guo Q, Pan WL, Li SQ, Li RY, Guo ZP, Song ZQ, Li SS, Dong XQ, Wang L, Fu R, Regnault P, Charef P, Mazur R, Patekar M. Secukinumab demonstrates high efficacy and a favorable safety profile over 52 weeks in Chinese patients with moderate to severe plaque psoriasis. Chin Med J (Engl). 2020 Nov 20;133(22):2665-2673. doi: 10.1097/CM9.0000000000001163. PMID 33060370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 664 patients were screened and 543 patients were randomized to one of three treatment groups in the induction period: secukinumab 300 mg (n=272), secukinumab 150 mg (n=136), and placebo (n=135)
Groups:
- Placebo: Placebo
- Placebo - Secukinumab 300mg: patients switched to AIN457 at week 12
Period: INDUCTION
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Placebo - Secukinumab 300mg
Started | 136 | 272 | 135 | 0
Completed | 134 | 270 | 133 | 0
Not Completed | 2 | 2 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0
Period: MAINTENANCE
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Placebo - Secukinumab 300mg
Started | 134 | 270 | 4 | 129
Completed | 127 | 266 | 2 | 126
Not Completed | 7 | 4 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 1
Period: OVERALL STUDY
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Placebo - Secukinumab 300mg
Started | 136 | 272 | 6 | 129
Completed | 126 | 264 | 2 | 124
Not Completed | 10 | 8 | 4 | 5
Not completed — Adverse Event | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Pregnancy | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 1 | 1 | 1
Not completed — discontinued follow up | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Total
Number analyzed (Participants) | 136 | 272 | 135 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.39) | 39.9 (12.35) | 40.1 (11.01) | 40.2 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 67 | 27 | 131
  Male | 99 | 205 | 108 | 412
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    East Asian | 109 | 220 | 109 | 438
    Southeast Asian | 19 | 32 | 16 | 67
    South Asian | 1 | 0 | 0 | 1
    West Asian | 0 | 3 | 0 | 3
    other | 6 | 17 | 10 | 33
    not reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Caucasian | 7 | 20 | 10 | 37
    Asian | 129 | 252 | 125 | 506

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) 75 (Multiple Imputation)
Description: Psoriasis Area and Severity Index (PASI) was assessed/calculated as per usual standard. result given in terms of count of participants with response in 100 imputations. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: Week 12
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo
Number analyzed (Participants) | 136 | 272 | 135
Participants | 112 | 254 | 6
Statistical Analysis 1: Comparison: Secukinumab 150mg vs Placebo; PASI 75; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 153.94, 95% CI 2-sided [54.02 to 438.67]
Statistical Analysis 2: Comparison: Secukinumab 300mg vs Placebo; PASI 75; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 557.98, 95% CI 2-sided [187.2 to 1663.4]

2. Primary Outcome: Investigator's Global Assessment (IGA) Mod 2011 0/1 (Multiple Imputation)
Description: Investigator assessed disease using a validated scale (IGA mod 2011) and rate the disease from a score of 0 (clear skin) to 4 (severe disease). result given in terms of count of participants with response in 100 imputations. The Investigator's Global Assessment (IGA) mod 2011 scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Treatment success was defined as achievement of IGA mod 2001 score of 0 or 1.
Time Frame: Week 12
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo
Number analyzed (Participants) | 136 | 272 | 135
Participants | 92 | 214 | 4
Statistical Analysis 1: Comparison: Secukinumab 150mg vs Placebo; IGA; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 75.82, 95% CI 2-sided [25.81 to 222.72]
Statistical Analysis 2: Comparison: Secukinumab 300mg vs Placebo; IGA; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 149.71, 95% CI 2-sided [51.83 to 432.42]

3. Secondary Outcome: Psoriasis Area and Severity Index (PASI) 90 (Multiple Imputation)
Description: as for outcome 1
Time Frame: Week 12
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo
Number analyzed (Participants) | 136 | 272 | 135
Participants | 85 | 210 | 2
Statistical Analysis 1: Comparison: Secukinumab 150mg vs Placebo; PASI 90; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 114.85, 95% CI 2-sided [26.94 to 489.59]
Statistical Analysis 2: Comparison: Secukinumab 300mg vs Placebo; PASI 90; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 246.12, 95% CI 2-sided [58.41 to 1037.1]

4. Secondary Outcome: Efficacy of Secukinumab in Maintaining PASI 75 Response at Week 52 in Subjects Who Were PASI 75 Responders at Week 12 (Multiple Imputation)
Description: as for outcome 1
Time Frame: Week 52
Population: full analysis set with measure
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg
Number analyzed (Participants) | 112 | 254
Participants | 94 | 235

5. Secondary Outcome: Efficacy of Secukinumab in Maintaining IGA Mod 2011 0 or 1 Response at Week 52 in Subjects Who Were IGA Mod 2011 0 or 1 Responders at Week 12 (Multiple Imputation)
Description: as for outcome 2
Time Frame: Week 52
Population: full analysis set with measure
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg
Number analyzed (Participants) | 92 | 214
Participants | 65 | 162

6. Secondary Outcome: PASI 50/75/90/100 and IGA Mod 2011 0 or 1 Response Over Time (Multiple Imputation)
Description: Number (%) of subjects with PASI 50, PASI 75, PASI 90, PASI 100 and IGA mod 2011 0 or 1 response
Time Frame: week 1, week 12, week 24, week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - AIN457 300 mg: patients switched to AIN457 at week 12
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Placebo - AIN457 300 mg
Number analyzed (Participants) | 136 | 272 | 135 | 129
Participants
  Week 1 IGA 0/1: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 1 IGA 0/1 | 0 | 1 | 0 | 0
  Week 1 PASI 50: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 1 PASI 50 | 5 | 25 | 1 | 0
  Week 1 PASI 75: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 1 PASI 75 | 0 | 0 | 0 | 0
  Week 1 PASI 90: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 1 PASI 90 | 0 | 0 | 0 | 0
  Week 1 PASI 100: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 1 PASI 100 | 0 | 0 | 0 | 0
  Week 12 IGA 0/1: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 12 IGA 0/1 | 92 | 214 | 4 | 0
  Week 12 PASI 50: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 12 PASI 50 | 130 | 267 | 16 | 0
  Week 12 PASI 75: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 12 PASI 75 | 112 | 254 | 6 | 0
  Week 12 PASI 90: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 12 PASI 90 | 85 | 210 | 2 | 0
  Week 12 PASI 100: number analyzed (Participants) | 136 | 272 | 135 | 0
  Week 12 PASI 100 | 28 | 81 | 1 | 0
  Week 16 IGA 0/1: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 16 IGA 0/1 | 100 | 219 | 2 | 32
  Week 16 PASI 50: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 16 PASI 50 | 134 | 270 | 4 | 108
  Week 16 PASI 75: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 16 PASI 75 | 124 | 261 | 3 | 72
  Week 16 PASI 90: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 16 PASI 90 | 98 | 233 | 2 | 22
  Week 16 PASI 100: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 16 PASI 100 | 39 | 99 | 0 | 3
  Week 24 IGA 0/1: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 24 IGA 0/1 | 91 | 217 | 1 | 88
  Week 24 PASI 50: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 24 PASI 50 | 135 | 271 | 4 | 123
  Week 24 PASI 75: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 24 PASI 75 | 123 | 257 | 2 | 113
  Week 24 PASI 90: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 24 PASI 90 | 93 | 230 | 2 | 94
  Week 24 PASI 100: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 24 PASI 100 | 47 | 107 | 0 | 31
  Week 52 IGA 0/1: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 52 IGA 0/1 | 79 | 194 | 0 | 96
  Week 52 PASI 50: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 52 PASI 50 | 128 | 269 | 4 | 126
  Week 52 PASI 75: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 52 PASI 75 | 111 | 259 | 4 | 119
  Week 52 PASI 90: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 52 PASI 90 | 86 | 218 | 1 | 101
  Week 52 PASI 100: number analyzed (Participants) | 136 | 272 | 4 | 129
  Week 52 PASI 100 | 42 | 110 | 1 | 55

7. Secondary Outcome: American Collage of Rheumatology (ACR) Response 20/50/70
Description: Percentage of patients who achieved ACR 20/50/70 at Week 12 and up to Week 52. The subset of patients who had active PsA at baseline included 7 patients in the secukinumab 150 mg group, 17 patients in the secukinumab 300 mg group and 4 patients in the placebo group. ACR 20, 50 or 70 responses correspond, respectively, to at least 20%, 50% or 70% improvement in comparison with baseline in the number of tender and swollen joint counts, in addition to similar improvements in at least three of five other measure of disability or disease activity
Time Frame: week 12, week 24, week 52
Population: full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150mg | Secukinumab 300mg | Placebo | Placebo - AIN457 300 mg
Number analyzed (Participants) | 7 | 17 | 4 | 4
Participants
  Week 12 ACR 20: number analyzed (Participants) | 7 | 16 | 4 | 0
  Week 12 ACR 20 | 4 | 13 | 0 | 0
  Week 12 ACR 50: number analyzed (Participants) | 7 | 16 | 4 | 0
  Week 12 ACR 50 | 3 | 12 | 0 | 0
  Week 12 ACR 70: number analyzed (Participants) | 7 | 16 | 4 | 0
  Week 12 ACR 70 | 2 | 6 | 0 | 0
  Week 24 ACR 20: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 24 ACR 20 | 5 | 14 | 0 | 2
  Week 24 ACR 50: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 24 ACR 50 | 4 | 10 | 0 | 1
  Week 24 ACR 70: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 24 ACR 70 | 2 | 6 | 0 | 1
  Week 52 ACR 20: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 52 ACR 20 | 4 | 13 | 0 | 3
  Week 52 ACR 50: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 52 ACR 50 | 3 | 11 | 0 | 2
  Week 52 ACR 70: number analyzed (Participants) | 7 | 16 | 0 | 4
  Week 52 ACR 70 | 2 | 8 | 0 | 0

8. Secondary Outcome: Time to PASI 75 Response up to Week 12
Description: as for outcome 1
Time Frame: week 12
Population: full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Secukinumab 150mg | Secukinumab 300mg
Number analyzed (Participants) | 136 | 272
days | 57 [51 to 57] | 55 [29 to 57]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Events and deaths occurring in this on-treatment period plus follow up (+30 days or +5 half- lives) are reported in the Adverse Event Information Tables.
Groups:
- AIN457 150 mg: AIN457 150 mg
- AIN457 300 mg: AIN457 300 mg
- Any AIN457 300 mg: Any AIN457 300 mg
- Any AIN457 Dose: Any AIN457 dose
Arm/Group | AIN457 150 mg | AIN457 300 mg | Any AIN457 300 mg | Any AIN457 Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/272 | 0/401 | 0/537 | 0/135
Serious Adverse Events (participants affected / at risk) | 5/136 | 9/272 | 14/401 | 19/537 | 2/135
Other Adverse Events (participants affected / at risk) | 115/136 | 221/272 | 312/401 | 427/537 | 71/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150 mg (N=136) | AIN457 300 mg (N=272) | Any AIN457 300 mg (N=401) | Any AIN457 Dose (N=537) | Placebo (N=135)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1 | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 2 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 150 mg (N=136) | AIN457 300 mg (N=272) | Any AIN457 300 mg (N=401) | Any AIN457 Dose (N=537) | Placebo (N=135)
Diarrhoea (Gastrointestinal disorders) | 13 | 31 | 42 | 55 | 12
Pyrexia (General disorders) | 4 | 14 | 18 | 22 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 9 | 18 | 22 | 31 | 4
Folliculitis (Infections and infestations) | 6 | 18 | 26 | 32 | 0
Influenza (Infections and infestations) | 17 | 28 | 38 | 55 | 4
Nasopharyngitis (Infections and infestations) | 15 | 44 | 57 | 72 | 5
Pharyngitis (Infections and infestations) | 14 | 24 | 35 | 49 | 7
Rhinitis (Infections and infestations) | 2 | 14 | 16 | 18 | 1
Tinea pedis (Infections and infestations) | 5 | 20 | 25 | 30 | 1
Tonsillitis (Infections and infestations) | 5 | 14 | 16 | 21 | 1
Upper respiratory tract infection (Infections and infestations) | 41 | 67 | 97 | 138 | 13
Blood uric acid increased (Investigations) | 4 | 4 | 6 | 10 | 5
C-reactive protein increased (Investigations) | 7 | 11 | 13 | 20 | 3
Gamma-glutamyltransferase increased (Investigations) | 2 | 10 | 12 | 14 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 2 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 11 | 22 | 23 | 34 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 25 | 56 | 76 | 101 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 12 | 16 | 3
Headache (Nervous system disorders) | 4 | 10 | 10 | 14 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 17 | 25 | 38 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 25 | 32 | 48 | 3
Eczema (Skin and subcutaneous tissue disorders) | 10 | 20 | 25 | 35 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 32 | 36 | 48 | 11
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 3 | 3 | 9 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 12 | 24 | 30 | 42 | 0
Hypertension (Vascular disorders) | 5 | 19 | 22 | 27 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03066609/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT03066609/SAP_001.pdf